CLINICAL TRIAL: NCT06235879
Title: Comparison Between Ultrasound Guided Pericapsular Nerve Group (PENG) Block and Interscalene Brachial Plexus Block for Postoperative Analgesia Following Shoulder Arthroscopy: Prospective, Randomized Controlled Trial
Brief Title: Comparison Between Pericapsular Nerve Group (PENG) Block and Interscalene Brachial Plexus Block for Postoperative Analgesia Following Shoulder Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Sabry B Mohamed, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD298/2023
Record Dates: First submitted 2024-01-20; First posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Pericapsular Nerve Block; Interscalene Brachial Plexus Block; Shoulder Arthroscopy
MeSH Terms: interventions — Control Groups; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control Group (Other): Patients will receive ultrasound guided Interscalene brachial plexus (ISB) block after induction of general anesthesia.
  Interventions: Other: Control Group (Interscalene brachial plexus block)
- Group B (Pericapsular nerve group (PENG) block) (Experimental): Patients will receive ultrasound guided Pericapsular nerve group (PENG) block after induction of general anesthesia
  Interventions: Procedure: Pericapsular nerve group (PENG) block

INTERVENTIONS:
Other: Control Group (Interscalene brachial plexus block) — Patients will receive ultrasound guided interscalene brachial plexus block after induction of general anesthesia.
  Scanning with SonoSite M-Turbo C ® Ultrasound device with HFL - 38 X Linear probe (Japan) with high frequency (6 -13 MHz) will be started just below the level of the cricoid cartilage medial to the sternocleidomastoid muscle.
  the transducer will be moved slightly laterally across the neck to identify the scalene muscles and the brachial plexus that is present between the anterior and middle scalene muscles at the level of the sixth cervical vertebra deep to the sternocleidomastoid muscle.
  The needle will be then inserted in-plane toward the brachial plexus, in a lateral-to-medial direction.
  After negative aspiration and assurance that high resistance to injection is absent, 0.25% bupivacaine hydrochloride will be injected in a 5-ml increment below the lower root, between the 3 roots, and above the upper root.(Total amount is 15 ml of 0.25% bupivacaine hydrochloride).
  Arms: Group A (Control Group
Procedure: Pericapsular nerve group (PENG) block — Patients will receive ultrasound guided Pericapsular nerve group (PENG) block after induction of general anesthesia.
  Using SonoSite M-Turbo C ® Ultrasound device with HFL - 38 X Linear probe (Japan) with high frequency (6 -13 MHz) ,A linear ultrasound probe will be placed longitudinally between the coracoid and the humeral head.
  After defining the humeral head, the tendon of the subscapular muscle and the deltoid muscle over it, a 50-mm needle will be inserted using the ''in plane'' technique. When the needle pass through the deltoid muscle and touched the subscapularis tendon, a bone-like hard tissue will be felt and the needle can't be advanced further.
  The needle tip will be placed between the deltoid muscle and subscapularis tendon, after a careful aspiration, 15 ml of 0.25% bupivacaine hydrochloride will be injected.
  Arms: Group B (Pericapsular nerve group (PENG) block)

SUMMARY:
The study aimed to compare ultrasound guided pericapsular nerve group (PENG) block versus interscalene brachial plexus block for postoperative analgesia following shoulder arthroscopy.

DETAILED DESCRIPTION:
Shoulder arthroscopy can effectively treat a number of injuries and diseases of the shoulder on an ambulatory basis. Although shoulder arthroscopy is considered minimally invasive, it is related to severe postoperative pain. The use of arthroscopy is popular because it decreases pain, shortens hospital stay, and improves patient satisfaction. However, immediate postoperative pain remains to be a problem in more than 40% of patients.

Regional anesthesia, especially peripheral nerve blocks have various advantages like decreased need for postoperative analgesics, decreased incidence of nausea and vomiting, shortened recovery time and hospital stay, Early ambulation and discharge.

Interscalene brachial plexus (ISB) block is considered the gold standard technique for pain management in shoulder surgery as it provides the most reliable analgesia. However, it has the potential for many complications. The most common of these complications is phrenic nerve palsy, which is reversible but may result in significant respiratory distress especially in patients with compromised respiratory function. Other less common yet serious complications include Horner's syndrome, recurrent laryngeal nerve block that may result in hoarseness of voice, vascular puncture, brachial plexus neuropathy, and unintended injection of local anesthetic into the subarachnoid space, epidural space, or vertebral artery.

Pericapsular nerve group (PENG) block is a new block that provides a pericapsular distribution with local anesthetic infiltration around the glenohumeral joint and provides analgesia by reaching the sensory nerve branches of the glenohumeral joint.

ELIGIBILITY:
Inclusion Criteria:

- Age from 18 to 60 years old. - Both genders. - BMI ≤35 kg/m2. - American Society of Anesthesiologists Physical Status (ASA-PS) Class I and II. - Patient who will be scheduled for an elective unilateral arthroscopic shoulder surgery.

Exclusion Criteria:

* Refusal of procedure or participation in the study
* Patient under age of 18 years old or above 60 years' old
* Physical status: ASA-PS III or above.
* Pregnancy or lactation.
* Infection at site of injection.
* Psychiatric illness.
* CNS Diseases like (epilepsy, stroke …etc.) or neurological disease affecting patient's upper limb.
* Evidence of coagulopathy or anticoagulation.
* Patients with respiratory disease, renal or hepatic insufficiency.
* infection of the skin in the puncture area.
* Allergy against any of the drugs to be used.
* Obesity (BMI >35 kg/m2).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
First time for requiring analgesia | 24 hours postoperatively
  First time for requiring analgesia. It will be defined as the time from recovery until VAS score greater than 3.

SECONDARY OUTCOMES:
Total amount of pethidine consumption in the first 24 hours | 24 hours postoperatively
  If the patient complained of pain, intravenous pethidine sulfate will be (50mg/dose) to be repeated on demand (VAS is > 3) provided that the total 24-hour dosage not to exceed 50 mg every 6 hours.
The degree of pain | 24 hours postoperatively
  The degree of pain will be measured using visual analogue scale (VAS)ranging from 0 to 10, where 0 no pain and 10 maximum pain. It will be evaluated on arrival to PACU (T0) then at 2, 4, 6, 12, and 24 h postoperatively.
Complications | 24 hours postoperatively
  Any complications during and after the performance of the block - for example, pneumothorax, Horner's syndrome, hoarseness of voice, difficulty in breathing, weakness, and paresthesia in the arm will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.